CLINICAL TRIAL: NCT01468103
Title: Laser Peripheral Iridotomy Versus Surgical Peripheral Iridectomy in Early Angle Closure:a Randomized Clinical Trial
Brief Title: Laser Iridotomy Versus Surgical Iridectomy in Early Angle Closure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Gao Xinbo, student, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19831105gaoxinbo
Record Dates: First submitted 2011-11-06; First posted 2011-11-09 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Intraocular Pressure Changes; Peripheral Anterior Synechiae Increasing
Keywords: intraocular pressure; Peripheral anterior synechiae

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PACS (Experimental): primary angle closure suspects
  Interventions: Procedure: Surgical Iridectomy; Procedure: Laser Iridotomy
- PAC (Experimental): primary angle closure
  Interventions: Procedure: Surgical Iridectomy; Procedure: Laser Iridotomy

INTERVENTIONS:
Procedure: Surgical Iridectomy — Surgical Iridectomy is now widely used in our clinical.
  Other Names: Peripheral Surgical Iridectomy
Procedure: Laser Iridotomy — alternative choice to surgical iridectomy
  Other Names: Peripheral Laser Iridotomy

SUMMARY:
This is a randomized controlled clinical trial to compare laser peripheral iridotomy(LPI) and surgical peripheral iridectomy. Subjects of primary angle closure suspect, primary angle closure will be randomized to undergo LPI or SPI. Subjects are proposed to be followed up for 3 years.

DETAILED DESCRIPTION:
The following will be studied:

1. To evaluate the safety of these two techniques for the treatment of angle closure.
2. To compare the anterior chamber reaction and IOP changes post surgery.
3. TO establish the UBM/ASOCT chamber angle parameters changes pre and post surgery.
4. To assess the development of PAS.

ELIGIBILITY:
Inclusion Criteria:

1. more than 50 years old
2. Diagnosis of either: Primary angle closure suspects, Primary angle closure in need of laser iridotomy or surgical iridectomy
3. Able to give Informed concent

Exclusion Criteria:

1. Ophthalmic diseases other than glaucoma and cataract
2. pseudophakic or aphakic patients
3. inability to attend regular follow-up assessment or to give informed written consent
4. Secondary causes of angle closure e.g. subluxed lens, uveitis, trauma and neovascular glaucoma
5. Participating in another study
6. monocular patients

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-08; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
intraocular pressure | 3 years

SECONDARY OUTCOMES:
Angle assessment parameters | 3 years
  Angle assessment parameters,such as anterior chamber openning distance,are acquired by anterior segment optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang X Lan, MD, Study Director — Sun Yat-sen University
Locations (1):
- ZhongShan Ophthalmic Center, Guangzhou, Guangdong, China